CLINICAL TRIAL: NCT01512615
Title: CopenHeart IE - A Randomized Clinical Trial Investigating the Effect and Meaning of Integrated Rehabilitation Versus Usual Follow-up of Patients Treated for Infective Endocarditis
Brief Title: CopenHeart IE - Integrated Rehabilitation of Patients Treated for Infective Endocarditis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Principal Investigator, Selina Kikkenborg Berg, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RHCopenHeartIE
Record Dates: First submitted 2012-01-11; First posted 2012-01-19 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Infective Endocarditis
Keywords: Rehabilitation; Exercise training; Psycho-educational care
MeSH Terms: conditions — Endocarditis | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Complex Cardiac Rehabilitation
  Interventions: Other: Complex Cardiac rehabilitation
- Control group (Experimental): Usual care
  Interventions: Other: Control group

INTERVENTIONS:
Other: Complex Cardiac rehabilitation — Complex Cardiac Rehabilitation consisting of exercise training (minimum 3 times a week for a total of twelve weeks) and psychoeducational care (5 sessions over 6 months)
  Arms: Intervention group
Other: Control group — Usual care, clinical control as provided by treating heart centre
  Arms: Control group

SUMMARY:
The aim of the study is to describe the effect and meaning of an integrated rehabilitation programme, consisting of physical training and psycho-educational care, for patients treated for infective endocarditis.

The hypothesis is, that integrated rehabilitation can improve mental health, physical capacity and other factors.

DETAILED DESCRIPTION:
Infective endocarditis (IE) is among the most serious infectious diseases in the western world. Treatment requires lengthy hospitalization, high dosage antibiotics and possible valve replacement surgery. Studies indicate that patients experience persisting physical symptoms, diminished quality of life and difficulties returning to work, up to a year post-discharge. No studies investigating the effect of, interventions aimed at relieving these problems, have been published.

A randomized clinical trial is conducted to investigate the effect and meaning of an integrated rehabilitation programme on the physical and psychosocial functioning of patients treated for IE. The trial is a multi-centre, parallel arm design. A mixed methods embedded experimental design is chosen to include both quantitative and qualitative data to evaluate the intervention. The intervention consists of five psycho-educational consultations provided by specialized nurses and a twelve week individualized exercise training programme provided by physiotherapists. A qualitative and a survey-based pre-study will be undertaken, to investigate post-discharge experiences and rehabilitation needs of patients treated for IE. A qualitative post-intervention study will explore rehabilitation participation experiences.

The hypothesis is, that integrated rehabilitation can improve mental health, physical capacity, self-rated health, quality of life, nutritional status, sleep-quality and body-image and reduce anxiety, depression, fatigue, health care utilisation, work cessation and mortality in patients treated for IE and that it is cost effective.

150 patients treated for leftsided- (native- or prosthetic valve) or cardiac device endocarditis will be included in the trial

Questionnaires, cardiopulmonary testing, 6 minute walking test and qualitative interviews will be used to evaluate the effect and meaning of the programme.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* treated for leftsided- (native- or prosthetic valve) or cardiac device endocarditis based on Duke Criteria
* 18 years or older
* speaking and understanding Danish
* providing written informed consent

Exclusion Criteria:

Patients:

* unable to understand study instructions
* with an ischemic event within the past 6 months
* who are pregnant or breastfeeding
* with reduced ability to follow the planned programme due to i.e. substance abuse problems or other somatic illness
* with considerable illness in the musculoskeletal system or with physical disability, which complicates exercise training
* whose physician advise against participation

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Mental component scale | 1, 4, 6 and 12 months
  Measured by the mental component scale (MCS) in the SF-36 questionnaire

SECONDARY OUTCOMES:
Change in physical capacity | 1, 4 and 6 months
  Measured by Peak VO2 via ergospirometry testing

CONTACTS AND LOCATIONS:
Overall Officials: Trine B Rasmussen, PhD fellow, Principal Investigator — Copenhagen University Hospital Rigshospitalet, University Hospital Gentofte; Selina K Berg, MScN, Ph.d., Principal Investigator — Copenhagen University Hospital Rigshospitalet, University Hospital Gentofte; Ann-Dorthe Zwisler, MD, Ph.d., Principal Investigator — Copenhagen University Hospital Rigshospitalet, National Institute of Public Health, University of Southern Denmark; Henning Bundgaard, MD, Ph.d., Principal Investigator — Rigshospitalet, Denmark; Philip Moons, Prof, PhD, Principal Investigator — Centre for Health Services and Nursing Research, KU Leuven-University of
Locations (1):
- Rigshospitalet / gentofte hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Rasmussen TB, Zwisler AD, Risom SS, Sibilitz KL, Christensen J, Bundgaard H, Moons P, Thygesen LC, Lindschou J, Norekval TM, Berg SK. Comprehensive cardiac rehabilitation for patients following infective endocarditis: results of the randomized CopenHeartIE trial. Eur J Cardiovasc Nurs. 2022 Apr 9;21(3):261-270. doi: 10.1093/eurjcn/zvab047. PMID 34089600
- [Derived] Rasmussen TB, Zwisler AD, Moons P, Berg SK. Insufficient living: experiences of recovery after infective endocarditis. J Cardiovasc Nurs. 2015 May-Jun;30(3):E11-9. doi: 10.1097/JCN.0000000000000144. PMID 24704921
- [Derived] Rasmussen TB, Zwisler AD, Sibilitz KL, Risom SS, Bundgaard H, Gluud C, Moons P, Winkel P, Thygesen LC, Hansen JL, Norekval TM, Berg SK; CopenHeartIE Group. A randomised clinical trial of comprehensive cardiac rehabilitation versus usual care for patients treated for infective endocarditis--the CopenHeartIE trial protocol. BMJ Open. 2012 Nov 21;2(6):e001929. doi: 10.1136/bmjopen-2012-001929. Print 2012. PMID 23175738